CLINICAL TRIAL: NCT01865630
Title: Phase I Safety, Blood Brain Barrier Permeability and Potential Efficacy of Etanercept for Aneurysmal Subarachnoid Hemorrhage
Brief Title: Safety and Efficacy Study of Etanercept for Aneurysmal Subarachnoid Hemorrhage
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI moved to another institution
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-3007-ETP
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Prophylactic treatment with Etanercept in aSAH.; Safety of Etanercept in the prevention of DCI in aSAH.
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Etanercept (Experimental): Patients with aneurysmal subarachnoid hemorrhage will be treated with etanercept, 25 mg subcutaneously starting within 36 hours of SAH, and then receive doses 3.5 days and 7 days later for a total of 3 doses.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Lyophilized powder for reconstitution/ 25 mg/vial. 25 mg subcutaneously starting within 36 hours of SAH, and then receive doses 3.5 days and 7 days later for a total of 3 doses.
  Other Names: Enbrel (Amgen Inc., CA)

SUMMARY:
Subarachnoid hemorrhage (SAH) is a special type of stroke that typically results from a ruptured intracranial aneurysm, a weakening in the wall of a blood vessel. This type of life-threatening bleeding occurs in over 3000 Canadians per year, usually in working age adults. Although this type of stroke accounts for only 5-10% of strokes, it contributes a disproportionately larger percent of overall stroke morbidity and mortality due in part to the young age of those affected. If one is fortunate enough to survive the initial bleeding episode and the subsequent surgical treatment of the aneurysm, a patient may still develop secondary strokes 3 to 14 days after the initial bleed. These delayed strokes are the most significant cause of morbidity and mortality after SAH and may be potentially preventable. Currently, there is only one medication (an anti-hypertensive) that has convincingly shown to improve outcomes after SAH. The molecular pathway causing these delayed strokes is still not clear, and this is an active area of research.

Animal studies have revealed that these delayed strokes may be caused by a pro-inflammation molecule called tumor necrosis factor alpha (TNFa). Delayed strokes were prevented experimentally by a TNFa blocker called etanercept. This clinical study, utilizing prophylactic treatment with etanercept in patients with SAH, will ensure the safety of this drug and determine its effectiveness in preventing delayed strokes.

DETAILED DESCRIPTION:
SAH from a ruptured cerebral aneurysm has an incidence of 10 per 100,000 Canadians (over 3000 people annually). If a person survives SAH from a ruptured intracranial aneurysm, the most common complication is delayed cerebral ischemia (DCI). This is the delayed neurologic deterioration associated with angiographic vasospasm. Vasospasm refers to the arterial constriction that typically begins 3 days after SAH, is maximal 7 to 8 days later and generally resolves by 14 days. About two-thirds of patients with SAH develop vasospasm, one-third develop DCI and one-sixth of SAH patients die or sustain permanent disability from DCI, despite aggressive medical/surgical intervention.

Nimodipine, a calcium-channel antagonist, is currently the only drug to convincingly improve outcomes after SAH. Randomized multi-centre clinical trials utilizing clazosentan, an endothelin receptor antagonist, demonstrated no change in clinical outcome despite significant decrease in large vessel vasospasm. These results have shifted the research in the pathophysiology of DCI to alternative mechanisms other than large vessel vasospasm.

It is known that the presence of blood in the subarachnoid space triggers massive local and systemic inflammation, including increase in the production of a pro-inflammatory cytokine called tumor necrosis factor alpha (TNFa). We have shown in mice that global, and smooth muscle-specific knockout of TNFa prevents increased myogenic tone and reduces brain injury after SAH. Furthermore, systemic or intrathecal treatment with etanercept may prevent the increase in myogenic tone observed after SAH and may reduce brain injury. Administration of etanercept to patients with SAH is a critical step in determining the safety and potential efficacy of TNFa antagonists in SAH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 75 years old.
* World Federation of Neurological Surgeons (WFNS) grade 2 to 4.
* Subarachnoid hemorrhage (SAH) on admission computed tomographic (CT) scan (diffuse clot present in both hemispheres or local thick SAH).
* Ruptured saccular aneurysm, confirmed by angiography (catheter or CT angiography [CTA]) and treated by neurosurgical clipping or endovascular coiling.
* External ventricular drain placed as part of routine care.
* Able to be dosed within 36 hours of injury
* Historical modified Rankin score of 0 or 1.
* Hemodynamically stable after resuscitation (systolic blood pressure [SBP] > 100 mm Hg).
* Aminotransferase levels no greater than twice the upper limit of normal, hemoglobin > 85 g/dL, platelets > 125,000 cells/mm3, serum creatinine < 177 μmol/L.
* Informed consent.

Exclusion Criteria:

* SAH due to causes other than saccular aneurysm (such as trauma or rupture of fusiform or infective aneurysm).
* Intraventricular or intracerebral hemorrhage, in the absence of SAH, or with only local, thin SAH.
* Angiographic vasospasm prior to clipping or endovascular procedure.
* Major complication during clipping or endovascular coiling, such as massive intraoperative hemorrhage, arterial occlusion or inability to clip or coil the ruptured aneurysm.
* Cardio-pulmonary resuscitation required following SAH.
* Women with a positive urine pregnancy test at screening.
* Body mass index > 35
* Severe or unstable concomitant condition or disease (e.g., known significant neurologic deficit, cancer, hematologic, or coronary disease), or chronic condition (e.g., psychiatric disorder), which, in the opinion of the investigator, would affect the assessment of the safety and tolerability of etanercept.
* Patients who have received an investigational product or participated in another clinical trial within 28 days prior to randomization or those who have already participated in the current study.
* History of hepatitis B or C, history of heart failure (etanercept may exacerbate heart failure), active infection or serious infection in the last 6 months, history of tuberculosis and history of malignancy, multiple sclerosis or history of seizures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Safety, blood brain barrier (BBB) permeability and potential efficacy of the TNFa antagonist, etanercept, in humans with subarachnoid hemorrhage (SAH). | Up to Week 12 post-SAH
  Phase 1 safety, feasibility study in which patients with aneurysmal subarachnoid hemorrhage (aSAH) will be treated with etanercept, 25 mg subcutaneously starting within 36 hours of SAH, then receive doses 3.5 days and 7 days later for a total of 3 doses. Patients must have the aneurysm secured by neurosurgical clipping or endovascular coiling and have an external ventricular drain placed as part of routine care. Other aspects of routine care include clinical monitoring (vital signs, neurological exam), daily bloodwork, daily cerebrospinal fluid (CSF) samples, and brain imaging typically magnetic resonance imaging/angiography (MRI/MRA) within 48 hours of coiling, and CTA at day 7-11 post-bleed. Etanercept levels determined by ELISA, will be measured in the blood and CSF samples, as well as IL-1 levels.
  Adverse events will be recorded in case-report forms. Total study duration for each patient is 12 weeks, including hospital stay and clinical follow-up at 4 and 12 weeks post-SAH.

SECONDARY OUTCOMES:
Pharmacokinetics (plasma and CSF concentrations) of etanercept by measuring daily plasma and CSF concentrations by enzyme-linked immunosorbent assay (ELISA). | Up to Week 12 post-subarachnoid hemorrhage
  Pharmacokinetic sampling to monitor plasma and cerebrospinal fluid levels of etanercept will be performed daily after first administration of etanercept until post-SAH day 14 or hospital discharge, whichever comes first.

OTHER OUTCOMES:
Serum biomarkers, radiologic and clinical outcomes. This is a composite outcome measure. | Up to Week 12 post-subarachnoid hemorrhage.
  * To measure biomarkers that may reflect the effects of etanercept, including plasma C reactive protein, plasma and CSF interleukin-1β (IL-1β) and white blood cell counts.
  * To determine radiologic outcomes as determined by angiographic vasospasm on computed tomographic angiograms (CTA), comparing baseline and 7 to 11 days after SAH, and cerebral infarctions on magnetic resonance imaging (MRI).This is standard of care performed within 48 hours of endovascular coiling and at 4-6 weeks).
  * To determine clinical outcome, assessed at 30 and 90 days after SAH using modified Rankin scale (mRS), extended Glasgow outcome scale (GOSe), telephone interview of cognitive status (TICS), dysexecutive questionnaire, and the Montreal cognitive assessment (MoCA).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Baker, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beeftink MM, Ruigrok YM, Rinkel GJ, van den Bergh WM. Relation of serum TNF-alpha and TNF-alpha genotype with delayed cerebral ischemia and outcome in subarachnoid hemorrhage. Neurocrit Care. 2011 Dec;15(3):405-9. doi: 10.1007/s12028-011-9556-1. PMID 21562930
- [Background] Gruber A, Rossler K, Graninger W, Donner A, Illievich MU, Czech T. Ventricular cerebrospinal fluid and serum concentrations of sTNFR-I, IL-1ra, and IL-6 after aneurysmal subarachnoid hemorrhage. J Neurosurg Anesthesiol. 2000 Oct;12(4):297-306. doi: 10.1097/00008506-200010000-00001. PMID 11147377
- [Background] Kerensky TA, Gottlieb AB, Yaniv S, Au SC. Etanercept: efficacy and safety for approved indications. Expert Opin Drug Saf. 2012 Jan;11(1):121-39. doi: 10.1517/14740338.2012.633509. Epub 2011 Nov 11. PMID 22074366
- [Background] Vecchione C, Frati A, Di Pardo A, Cifelli G, Carnevale D, Gentile MT, Carangi R, Landolfi A, Carullo P, Bettarini U, Antenucci G, Mascio G, Busceti CL, Notte A, Maffei A, Cantore GP, Lembo G. Tumor necrosis factor-alpha mediates hemolysis-induced vasoconstriction and the cerebral vasospasm evoked by subarachnoid hemorrhage. Hypertension. 2009 Jul;54(1):150-6. doi: 10.1161/HYPERTENSIONAHA.108.128124. Epub 2009 May 26. PMID 19470883
- [Background] Zhou QH, Sumbria R, Hui EK, Lu JZ, Boado RJ, Pardridge WM. Neuroprotection with a brain-penetrating biologic tumor necrosis factor inhibitor. J Pharmacol Exp Ther. 2011 Nov;339(2):618-23. doi: 10.1124/jpet.111.185876. Epub 2011 Aug 10. PMID 21831964